CLINICAL TRIAL: NCT03451916
Title: Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study, Designed to Determine the Efficacy, Safety, and Tolerability of Intramuscular Administration of Allogeneic PLX-PAD Cells for the Treatment of Muscle Injury Following Arthroplasty for Hip Fracture
Brief Title: Treatment of Muscle Injury Following Arthroplasty for Hip Fracture (HF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pluristem Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: PLX-HF-01
Record Dates: First submitted 2018-02-25; First posted 2018-03-02 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Hip Fracture
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Intervention Model Description: , subjects will be randomized using a 1:1 allocation scheme to either 150×10^6 PLX-PAD cells or to placebo treatment, respectively
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PLX-PAD (Experimental): • Arm 1 - PLX-PAD (120 subjects): 150×10^6 PLX-PAD cells (10×10^6 cells/mL) in a mixture containing 10% DMSO (v/v), 5% HSA (w/v) and PlasmaLyte.
  Interventions: Drug: PLX-PAD
- Placebo (Placebo Comparator): Arm 2 Placebo (120 subjects): Placebo (solution comprised of 10% DMSO [v/v], 5% HSA [w/v], and PlasmaLyte, without cells).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PLX-PAD — PLX-PAD (120 subjects): 150×10^6 PLX-PAD cells (10×10^6 cells/mL) in a mixture containing 10% DMSO (v/v), 5% HSA (w/v) and PlasmaLyte
  Arms: PLX-PAD
Drug: Placebo — Arm 2 Placebo (120 subjects): Placebo (solution comprised of 10% DMSO [v/v], 5% HSA [w/v], and PlasmaLyte, without cells).
  Arms: Placebo

SUMMARY:
The objectives of this study are to assess the efficacy, safety, and tolerability of PLX-PAD intramuscular administration for the treatment of muscle injury following arthroplasty for HF.

DETAILED DESCRIPTION:
This will be a Phase III, multinational, randomized, double-blind, placebo-controlled study, assessing the efficacy, safety, and tolerability of intramuscular (IM) administration of allogeneic PLX-PAD cells for the treatment of muscle injury following arthroplasty for HF as compared to placebo treatment. Both treatment arms will receive standard of care treatment per local practice.

The study will comprise 2 periods:

1. Main study period - from Screening to 52 weeks post-treatment. During this period, the subjects will have the following study visits: Screening, Day 0 (treatment and surgery day), Day 1, Day 5, Week 6, Week 12, Week 26 and Week 52.
2. Safety follow-up period - from Week 52 to Week 104. During this safety follow-up period, there will be a phone call visit at Week 104 and Only survival and quality of life data, serious adverse events (SAEs) and new malignancy adverse events will be collected.

The main study period will comprise 4 periods:

1. Screening and pre-surgery time
2. Surgery and treatment with PLX-PAD or placebo (Day 0)
3. Hospital follow-up until Day 5±1, at least
4. Follow-up period up to 52 weeks following study treatment administration. Subjects will be assessed for study eligibility before the emergency surgery for HF. After being found eligible, subjects will be randomized using a 1:1 allocation scheme to either 150×106 PLX-PAD cells or to placebo treatment, respectively. Within 48 hours of admission and up to 72 hours following fracture, subjects will undergo HA or THA. During the surgical procedure, the subjects will receive the investigational product in accordance with the treatment group to which they were randomized. Thereafter, visits will be conducted at Days 1 and 5±1, and at Weeks 6, 12, 26, 52 and 104.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects
2. Subjects up to 90 years of age, inclusive, at the time of Screening
3. Subjects suffering low energy trauma with intracapsular neck of femur fracture.
4. Planned to be treated with total hip arthroplasty (THA) or hemi-arthroplasty (HA) within 48 hours of hospital admission and 72 hours post fracture.
5. Subjects able to walk 10 feet/3 meters before the fracture.
6. Signed an informed consent.

Exclusion Criteria:

* 1. Any significant musculoskeletal, neurologic or neuromuscular disease causing muscle weakness and/or affecting mobility 2. Current fracture is due to bone pathology other than osteoporosis or due to major trauma 3. Planned orthopedic surgery on lower limbs (excluding hip arthroplasty) within the next 12 months.

  4. Diabetes mellitus with HbA1c >10% at Screening. 5. Known current or history of proliferative retinopathy or diabetic retinopathy.

  6. Known active Hepatitis B virus or Hepatitis C virus infection. 7. Known human immunodeficiency virus (HIV) infection, severe uncontrolled inflammatory disease or severe uncontrolled autoimmune disease (e.g., ulcerative colitis, Crohn's disease, etc).

  8. Subjects on renal replacement therapy or with estimated glomerular filtration rate (eGFR) <15 mL/min/1.73m2 9. Severe congestive heart failure symptoms (New York Heart Association [NYHA] Stage IV).

  10. Known uncontrolled severe hypertension. 11. Treatment with anabolic steroids within 6 months prior to study start 12. Active malignancy or history of malignancy within 3 years prior to study start 13. Known moderate to severe dementia or severe psychiatric disorder. 14. Known allergies to any of the following: dimethyl sulfoxide (DMSO), human serum albumin (HSA), bovine serum albumin, PlasmaLyte.

  15. History of allergic/hypersensitivity reaction to any substance having required hospitalization and/or treatment with IV steroids/epinephrine 16. Pulmonary disease requiring supplemental oxygen treatment on a daily basis. 17. life expectancy of less than 6 months, for reasons other than HF complications, 18. Subject is currently enrolled in or has not yet completed a period of at least 30 days since ending other investigational device or drug trial(s).

  19. In the opinion of the Investigator, the subject is unsuitable for participating in the study.

Ages: 0 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2023-09-06 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB) score | Week 26.

SECONDARY OUTCOMES:
Hip abduction strength of the injured leg | Week 26.
Change from baseline to Week 52 in lower extremity measure (LEM) (retrospective collection of pre-fracture LEM at Day 5±1). | baseline to Week 52
SPPB score | Week 52.
  The Short Physical Performance Battery (SPPB) is an objective assessment tool for evaluating lower extremities function. The SPPB consists of 3 types of physical maneuvers: balance test, speed gait test, and chair stand test. Results from each maneuvers test are scored on a scale of 0 to 4, with an increasing composite score indicating an improved lower extremities function level. The total maximum score of SPPB is 12.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (3):
  - University Of California Davis,4860 Y Street, Sacramento, California
  - Denver Metro Orthopedics, P.C. 499 E. Hampden Avenue, Suite 140 Englewood, CO 80113, Denver, Colorado
  - ANTRIA, INC,300 Indian Springs Road,Indiana, Indiana, Pennsylvania
- Bulgaria (4):
  - MHAT "Ljulin" Department of Orthopedy and Traumatology, Sofia
  - MHAT "Serdika" Department of Orthopedy and Traumatology, Sofia
  - Military Medical Academy, Sofia
  - Specialized Hospital for Active Treatment in Orthopedy, Sofia
- Germany (3):
  - Charite - Campus Mitte,Campus Virchow-Klinikum, Berlin
  - Universitaetsklinikum Carl Gustav Carus an der Technischen Universitaet Dresden, Dresden
  - Universitaetsklinikum Muenster, Münster
- Israel (6):
  - Carmel Medical Center,7 Michal St, Haifa
  - Shaare Zedek Medical Center,The Orthopedic Department,Shmu'el Bait St. 12, Jerusalem
  - Meir Medical Center-Internal Medicine E;59 Tshernichovsky Street, Kfar Saba
  - The Chaim Sheba Medical Center,Tel Hashomer, Ramat Gan
  - Kaplan Medical Center,Pasternak St., P.O.B 1,Rehovot, Rehovot
  - Sourasky Medical Center,6 Weizmann St; Harrison Building 6 Floor, Tel Aviv
- John Radcliffe Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No